CLINICAL TRIAL: NCT01274780
Title: Metabolic Effects of Atazanavir/Ritonavir Versus Darunavir/Ritonavir in Combination With Tenofovir/Emtricitabine in naïve HIV-1 Infected Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Juan A. Arnaiz (Other)
Responsible Party: Sponsor-Investigator, Juan A. Arnaiz, Clinical research Manager, Hospital Clinic of Barcelona
Organization: Hospital Clinic of Barcelona (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATADAR
Record Dates: First submitted 2011-01-11; First posted 2011-01-12 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: HIV-1
MeSH Terms: interventions — Darunavir; Ritonavir; Tenofovir; Emtricitabine; Atazanavir Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Darunavir / Ritonavir (Experimental)
  Interventions: Drug: Darunavir / Ritonavir + Tenofovir / Emtricitabine
- Atazanavir / Ritonavir (Experimental)
  Interventions: Drug: Atazanavir / Ritonavir + Tenofovir / Emtricitabine

INTERVENTIONS:
Drug: Darunavir / Ritonavir + Tenofovir / Emtricitabine — oral, 800/100 mg, qd + oral, 300/200 mg, qd
  Arms: Darunavir / Ritonavir
Drug: Atazanavir / Ritonavir + Tenofovir / Emtricitabine — oral, 300/100 mg, qd + oral, 300/200 mg, qd
  Arms: Atazanavir / Ritonavir

SUMMARY:
This is a prospective, open controlled trial in which naïve HIV-1 patients will be randomized to receive atazanavir / ritonavir or darunavir / ritonavir in combination with tenofovir / emtricitabine. They will be followed up during 96 weeks to determinate the cholesterol levels.

Randomization will be stratified according to the values of the ratio of total cholesterol/HDL cholesterol obtained during the screening visit (as they will be <4.5 or ≥ 4.5).

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both sexes aged 18 years or more. Women of childbearing potential must commit to sexual abstinence or use barrier contraceptive methods during the study.
2. Diagnosis of infection by HIV-1 (according to standard diagnostic criteria)
3. Not previously treated with antiretroviral drugs
4. Plasma viral load > = 1000 copies / ml
5. Clinically stable patients in the investigator's opinion at the time of inclusion
6. Able to meet the schedule of study visits and other protocol requirements
7. Written informed consent to participate in the study and undergo tests and examinations that entails

Exclusion Criteria:

1. ALT, AST levels greater than or equal to 5 times ULN (upper limit of normal)
2. serum creatinine level greater than 2 times ULN
3. Diabetes Mellitus (according to clinical and / or use of anti-diabetic agents)
4. Obesity (BMI ≥ 30 kg/m2)
5. Use of drugs that may affect lipid and / or glucose metabolism for at least 30 days prior to inclusion in the study.
6. Active opportunistic infection requiring intravenous treatment
7. Patients with known hypersensitivity to any of the products under study
8. Use of drugs formally contraindicated in the product information for any of the drugs under study
9. Contraindication to the use of any of the drugs under study
10. Women pregnant or lactating at the time of study inclusion or anticipating pregnancy in the follow-up period provided by the test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2011-05; Primary Completion 2013-05 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Changes in total cholesterol | 24 weeks

SECONDARY OUTCOMES:
Blood levels of: triglycerides, total cholesterol, LDL cholesterol, HDL cholesterol and ratio of total cholesterol/HDL cholesterol | 24, 48 and 96 weeks
Cardiovascular risk according to the Framingham scale. | 24, 48 and 96 weeks.
Glycemic profile (including glucose, insulin and HOMA (homeostatic model assessment index)) | 24, 48 and 96 weeks
inflammatory markers (protein C-reactive protein and interleukin-6) and anti-inflammatory (adiponectin) | 24, 48 and 96 weeks
RNA viral load <50 copies / mL | 24, 48 and 96 weeks.
CD4+ cells count | 24, 48 and 96 weeks
clinical adverse events, including events related to depositional patterns, laboratory abnormalities and incidence of treatment discontinuation because of toxicity or intolerance in each of the treatment arms. | 24, 48 and 96 weeks
distribution of body fat by DEXA (X-ray densitometry dual energy level) and CT (Computerized Axial Tomography)scan | 48 and 96 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Gonzalez-Cordon A, Domenech M, Camafort M, Martinez-Rebollar M, Torres B, Laguno M, Rojas J, Lonca M, Blanco JL, Mallolas J, Gatell JM, de Lazzari E, Martinez E. Subclinical cardiovascular disease in patients starting contemporary protease inhibitors. HIV Med. 2018 May 10. doi: 10.1111/hiv.12619. Online ahead of print. PMID 29745457
- [Derived] Martinez E, Gonzalez-Cordon A, Ferrer E, Domingo P, Negredo E, Gutierrez F, Portilla J, Curran A, Podzamczer D, Ribera E, Murillas J, Bernardino JI, Santos I, Carton JA, Peraire J, Pich J, Deulofeu R, Perez I, Gatell JM; ATADAR Study Group. Differential body composition effects of protease inhibitors recommended for initial treatment of HIV infection: a randomized clinical trial. Clin Infect Dis. 2015 Mar 1;60(5):811-20. doi: 10.1093/cid/ciu898. Epub 2014 Nov 10. PMID 25389256
- [Derived] Martinez E, Gonzalez-Cordon A, Ferrer E, Domingo P, Negredo E, Gutierrez F, Portilla J, Curran A, Podzamczer D, Murillas J, Bernardino JI, Santos I, Carton JA, Peraire J, Pich J, Perez I, Gatell JM; ATADAR Study Group. Early lipid changes with atazanavir/ritonavir or darunavir/ritonavir. HIV Med. 2014 Jul;15(6):330-8. doi: 10.1111/hiv.12121. Epub 2014 Jan 12. PMID 24417772